CLINICAL TRIAL: NCT05585281
Title: A Prospective, Single-Arm, Single-Center, Phase II Clinical Trial Evaluating the Efficacy and Safety of Fluzoparib Combined With QL1101 for Maintenance Treatment in Patients With Advanced Epithelial Ovarian Cancer Following Response After First-line Platinum-containing Chemotherapy
Brief Title: A Study of Fluzoparib Combined With QL1101 Maintenance Treatment in Patients With Advanced Ovarian Cancer Following Response on Front-Line Platinum-Based Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yongpeng Wang (Other)
Responsible Party: Sponsor-Investigator, Yongpeng Wang, Principal Investigator, Liaoning Cancer Hospital & Institute
Organization: Liaoning Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220501
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving Fluzoparib+ QL1101 (Experimental): Participants will be administered QL1101 7.5 milligram per kilogram (mg/kg) via a 30 minute (min) intravenous (IV) infusion on Day 1 of each 21-day cycle. Fluzoparib will be administered orally twice daily continuously throughout each 21-day cycle. On Day 1 of each cycle, fluzoparib will be administered upon completion of QL1101 infusion. The starting dose of fluzoparib will be based on the participant's Baseline actual body weight or platelet count.
  Interventions: Drug: Fluzoparib; Biological: QL1101

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib Orally twice daily
Biological: QL1101 — Maintenance QL1101 7.5 mg/kg will be administered via a 30-minute IV infusion on Day 1 of every 21-day cycle in the absence of progressive disease (PD), unacceptable toxicity, participant withdrawal, Investigator's decision, or death. QL1101 will be administered for up to 10 months during the maintenance phase or up to a total of 15 months inclusive of approximately 5 months of QL1101 received with chemotherapy.

SUMMARY:
This is a Prospective,Single-Center, Single-Arm, Phase 2 study to evaluate the efficacy and safety of Fluzoparib Combined With QL1101, as maintenance treatment, in patients with Advanced FIGO Stage III or IV High Grade Serous or Endometrioid Ovarian, Fallopian Tube, or primary peritoneal cancer following front-line platinum-based chemotherapy with QL1101. Eligible participants who achieve complete response (CR) or partial response (PR) following treatment with platinum-based chemotherapy in addition to QL1101 will be enrolled in the study and will receive maintenance treatment with fluzoparib (for up to 2 years) combined with QL1101 (for up to 10 months during the maintenance phase or up to a total of 15 months inclusive of the approximately 5 months of bevacizumab received with chemotherapy) or until disease progression, unacceptable toxicity, participant withdrawal, Investigator's decision, or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

I-1.Patients voluntarily participated in this study and signed the informed consent.

I-2.Age 18-70 years, female. I-3.Eastern Cooperative Oncology Group (ECOG) performance status 0-1. I-4.Patients with newly diagnosed, histologically confirmed, high grade serous or high grade endometrioid ovarian cancer, fallopian-tube cancer, or primary peritoneal cancer（FIGO Stage III or IV）.

I-5.Completion of ideal tumor cytoreduction (either intermediate cytoreduction or initial cytoreduction).

I-6.First line therapy with platinum-taxane chemotherapy consists of a minimum of 6 treatment cycles and a maximum of 8 treatment cycles in patients who have achieved complete response (CR) or partial response (PR).

I-7.Patients who must receive at least 4 cycles of platinum-based therapy if non-hematologic toxicity specifically associated with platinum-based therapy (i.e., neurotoxicity, hypersensitivity reactions, etc.) necessitates early termination.

I-8.Those who can swallow tablets normally.

I-9.The functions of vital organs meet the following requirements:

1. Absolute neutrophil count ≥ 1.5 × 109/L;
2. Platelets ≥ 90 × 109/L;
3. Hemoglobin ≥ 100 g/L;
4. Serum albumin ≥ 30 g/L;
5. Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN);
6. ALT and AST ≤ 3 × ULN; in case of liver metastases, ALT and AST < 5 × ULN;
7. Serum creatinine ≤ 1.5 × ULN;
8. International normalized ratio (INR) ≤1.5 and activated prothrombin time (aptt) ≤1.5× ULN in patients not receiving anticoagulants.

I-10.Maintenance therapy is initiated within 8 weeks, counting from the last day of the last chemotherapy session, and all major toxicities from prior chemotherapy must be resolved by maintenance therapy to CTC Adverse Event grade 1 or better (except alopecia and peripheral neuropathy).

I-11.Normal blood pressure or adequately treated and controlled hypertension (systolic blood pressure ≤ 140 mmHg and/or diastolic blood pressure ≤ 90 mmHg) .

I-12.Willingness to undergo genetic testing: including germline and/or systemic BRCA1/2 testing, HRD testing, etc.

I-13.Non-surgical sterilization or female patients of childbearing age need to use two medically approved contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study treatment period and within 3 months after the end of the study treatment period; non-surgical sterilized female patients of childbearing age must have a negative serum human chorionic gonadotropin(HCG) test within 72 hours before the first dose, and must be non-lactating; for male patients whose partners are women of childbearing age, two effective methods of contraception should be used during the study treatment period and for 3 months after the end of the study treatment period.

Exclusion Criteria:

E-1.Non-epithelial origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors).

E-2.Ovarian tumors of low malignant potential (e.g. borderline tumors), or mucinous carcinoma.

E-3.Clinical evidence of stable disease or progressive disease following treatment at the end of the first-line chemotherapy.

E-4.Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS)Patients with a history of localized malignancy diagnosed over 5 years ago, who have completed all treatment and have no recurrent or metastatic disease prior to enrollment may be enrolled.

E-5.Patients with myelodysplastic syndrome/acute myeloid leukemia history. E-6.Patients receiving radiotherapy within 6 weeks or Major surgery within 4 weeks prior to study treatment.

E-7.Any previous treatment with PARP inhibitor, including fluzoparib. E-8.Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.

E-9.Clinically significant (e.g. active) cardiovascular disease, including:

1. New York Heart Association (NYHA) grade 2 or higher heart failure.
2. Unstable angina pectoris.
3. Myocardial infarction within 1 year.
4. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.
5. Qtc>470ms. E-10.Patients who underwent cytoreductive surgery more than once before maintenance treatment（Patients who were considered unresectable at diagnosis only received biopsy or ovarian resection, and then continued chemotherapy for intermediate cytoreductive surgery may be enrolled）.

E-11.Patients who have received chemotherapy for abdominal or pelvic tumors, including those who received chemotherapy for early diagnosis of ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

E-12.Patients with synchronous primary endometrial cancer unless both of the following two criteria are met:

1. Sage < 2.
2. Less than 60 years old at the time of diagnosis of endometrial cancer with stage ia or ib grade 1 or 2, or stage ia grade 3 endometrioid adenocarcinoma or ≥ 60 years old at the time of diagnosis of endometrial cancer with stage ia grade 1 or 2 endometrioid adenocarcinoma. Patients with serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium are not eligible.

E-13.Pregnant or lactating women. E-14.Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin, and nelfinavir.

E-15.History of allergic reactions to carboplatin. E-16.Participation in another clinical study with an investigational product.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-27 (Estimated); Primary Completion 2025-11-07 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival(PFS) | up to 2 years
  PFS by investigator's assessment

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up. For subjects who survived or were lost to follow-up by the data analysis cutoff date, survival was truncated by the subject's last known survival time.
Second Progression Free Survival（PFS2） | up to 2 years
  Time to progression on the next anticancer therapy (PFS2) From date of start of next anticancer therapy to date of first documented progression of date of death from any cause, whichever comes first. The impact of this study's maintenance regimen on patient follow-up was determined by assessing the time from enrollment to second progression (PFS2), or the purpose of the PFS2 analysis was to demonstrate whether maintenance treatment could reduce the benefit provided by follow-up.
Time to start of first subsequent therapy or death（TFST） | up to 2 years
  The evaluation of the efficacy of first-line platinum-based chemotherapy and maintenance therapy by assessing the time to first follow-up or death, in addition to the similar assessment role as for PFS, allows evaluation of whether the regimen has an impact on follow-up and, if follow-up is delayed, on PFS2 and OS.
Health-related quality of life（HRQoL） | up to week 24
  To evaluate the effects of this trial protocol on health-related quality of life (HRQoL) in patients with high-risk advanced epithelial ovarian cancer as assessed by the Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy-Ovary (FACT-O).The TOI ranges from 0 to 100, with higher scores associated with higher HRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Yongpeng Wang, Shenyang, China